CLINICAL TRIAL: NCT06226038
Title: Effect of the Modified Magnetic Interim Denture on Dental Implant Stability and Marginal Bone Level: a Double-blind Randomized Controlled Trial Study
Brief Title: Effect of Static Magnetic Field on Dental Implant Stability.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: COA. MURA2023/919
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Implant Site Reaction
Keywords: Static magnetic field; Dental implant; Bone healing
MeSH Terms: interventions — Stainless Steel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With magnet (Experimental)
  Interventions: Other: Magnet disc
- Without magnet (Sham Comparator)
  Interventions: Other: Stainless steel

INTERVENTIONS:
Other: Magnet disc — Magnetic field promote proliferation and stimulate osteoblast differentiation
  Arms: With magnet
Other: Stainless steel — For control
  Arms: Without magnet

SUMMARY:
To evaluate the effect of static magnetic field on dental implant to bone integration.

DETAILED DESCRIPTION:
Bone to implant integration depend on bone healing. Magnetic field was proved to promote and make bone to implant integration happen faster. We decided to investigate by placing 2 dental implants in lower jaw of complete edentulous patients with specialised temporary dentures. Said denture will have neodymium magnet on one side, completely embedded in acrylic mass.

ELIGIBILITY:
Inclusion Criteria:

* healthy, complete edentulous area

Exclusion Criteria:

* uncontrolled NCDs patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant stability quotient | 90 days
  Stability quantity of dental implant measured by resonance frequency analysis machine

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol university, Bangkok, Payatai, Thailand

IPD SHARING:
Plan to Share IPD: No